CLINICAL TRIAL: NCT06395844
Title: Safety and Efficacy of Intraperitoneal Injection of METR-NK Cells as Neoadjuvant Therapy for Advanced Epithelial Ovarian Cancer: A Single-arm, Single-center, Exploratory Clinical Study
Brief Title: Safety and Efficacy of Intraperitoneal Injection of METR-NK Cells as Neoadjuvant Therapy for Advanced Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Collaborators: Anhui Kecheng intelligent health technology Co., LTD (Unknown)
Responsible Party: Principal Investigator, Bai-Rong Xia, Director of Gynecological Surgery, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 No. 050
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- METR-NK cell（metabolic remodeling nature killer cells） (Experimental): Intraperitoneal allogeneic METR-NK cells infusion ： Dilute 200 mL of METR-NK cells in 1500 mL of 0.9% saline solution at 37°C. The minimum amount of METR-NK cells infused each time should be no less than 7.5×10^7 cells per kilogram. Continuous infusion for 2 days constitutes one course, with 4 courses, with 13-day interval between each course
  Interventions: Drug: METR-NK cell(Metabolic Remodeling Nature Killer Cells)

INTERVENTIONS:
Drug: METR-NK cell(Metabolic Remodeling Nature Killer Cells) — The minimum amount of METR-NK cells infused each time should be no less than 7.5×10^7 cells, Continuous infusion for 2 days constitutes one course, with 4 courses. The infusion is given every 2 weeks.

SUMMARY:
The goal of this type of clinical trial study is to evaluate the safety and efficacy of metabolic remodeling nature killer cells as neoadjuvant therapy in newly diagnosed patients with advanced ovarian cancer

DETAILED DESCRIPTION:
Peripheral blood will be collected from a vein of arm. Peripheral blood mononuclear cells (PBMc) will be isolated and purified for NK manufacturing. The addition of key metabolic molecules in the medium remodeled the metabolic network of NK cells, significantly reduced the aging phenomenon of NK cells in the culture process, improved the cell activity of NK cells and enhanced the cytotoxicity of NK cells. After 14 days cultivation, activated METR-NK will be harvested and formulated for clinical administration.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old (≥18, ≤70);
* Open surgery, laparoscopic surgery, or coarse needle biopsy for histopathological confirmation of advanced (FIGO IIIC/IV stage) high-grade serous ovarian cancer, high-grade endometrioid carcinoma, primary peritoneal carcinoma, and/or fallopian tube carcinoma, etc.;
* ECOG score: 0-1;
* Blood and tissue specimens before, during, and after treatment can be obtained, and subjects agree to submit blood and tissue specimens to the central laboratory for the purpose of expanding research in this trial;
* At least one lesion measurable by CT/MRI according to RECIST 1.1 criteria;
* Expected survival of at least 3 months;
* Patients judged by professional gynecologic oncologists as unable to achieve R0 resection or intolerant to surgery.

  * Criteria for determining inability to achieve R0 resection include but are not limited to: Fagotti laparoscopic score ≥8 points; When laparoscopic evaluation is difficult to implement, an upper abdominal CT score ≥3 points may be used;
  * Criteria for intolerance to surgery may include: Advanced age: age ≥70; Body mass index: BMI ≥40.0; Multiple chronic diseases; Malnutrition or hypoalbuminemia; Moderate to large amount of ascites; Newly diagnosed venous thromboembolism (survival period greater than 12 weeks);
* Major organ function meets the following criteria within 7 days before treatment: Hematological examination: Hemoglobin ≥90g/L, white blood cell count ≥3×10^9/L, absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥90×10^9/L; Kidney: Serum creatinine <1.5 mg/dL, glomerular filtration rate (GFR) ≥50 ml/min (based on the Fairview Laboratories formula at screening); Liver: AST, ALT, and alkaline phosphatase <3 times the upper limit of normal for the institution, total bilirubin <1.5 times the upper limit of normal for the institution; Lung function: Resting oxygen saturation ≥90%; Cardiac function: Left ventricular ejection fraction (LVEF) ≥40% by echocardiography, MUGA, or cardiac MRI; no evidence of uncontrolled angina, severe uncontrolled ventricular arrhythmias, or acute ischemia or active conduction system abnormalities on electrocardiography;
* No history of intestinal obstruction within two months;
* Reproductive-age patients must take effective contraceptive measures;
* Subjects voluntarily join this study and sign an informed consent form (ICF);
* Good compliance is expected, and subjects are able to follow up on efficacy and adverse reactions as required by the protocol.

Exclusion Criteria:

* Patients who have received drugs or other cell immunotherapy in other clinical trials within 28 days before the screening period;
* Patients who have had other malignant tumors in the past 5 years;
* Acute illnesses are ongoing, or severe illnesses have occurred in the past 2 years, such as patients with active infections or fever, cardiovascular diseases (Grade III or IV heart failure), mental health issues (such as alcoholism, drug abuse);
* History of immunodeficiency, including HIV-positive status or other acquired, congenital immunodeficiency diseases;
* Organ transplant or organ failure patients, patients receiving immunosuppressive therapy after organ transplantation, or patients taking immunosuppressive drugs long-term;
* Thromboembolic events such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism within 6 months;
* Known allergy to any component of the final product of METR-NK preparation, including human serum albumin;
* Breastfeeding during the screening period or female subjects with positive serum or urine pregnancy tests;
* Patients with mental illnesses, including epilepsy, dementia, severe depression, bipolar disorder, etc.;
* Other conditions deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3-month
  the percentage of patients received R0 resection after METR-NK cells as neoadjuvant therapy for advanced epithelial ovarian cancer

SECONDARY OUTCOMES:
Overall Response Rate (ORR) After Neoadjuvant treatment | 3-month
  Overall Response Rate according to RECIST1.1 after Neoadjuvant treatment. ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Pathological complete remission rate | 3-month
  No residual invasive carcinoma was found under the microscope, but ductal carcinoma in situ could be found; In addition, compare the amount of cancer cells in the specimen before and after the new adjuvant therapy, and use of the Miller Payne grading system to evaluate the effect of the new adjuvant therapy
Disease control rate | 3-month
  the percentage of patients with complete response, partial response, and stable disease for more than 4 weeks in which response can be evaluated
Progression free survival | 2-years
  the date of enrollment to the date of the first onset of disease progression or death from any cause, whichever comes first
Survival rate | 3-years
  the date of enrollment to the date of death from any cause
Adverse event | 3-month
  Adverse medical events in clinical trial subjects treated with METR-NK cells

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Cancer Hospital, Hefei, Anhui, China